CLINICAL TRIAL: NCT02599298
Title: Sleep Study-Guided Multidisciplinary Therapy for Patients Presenting With Acute Coronary Syndrome
Acronym: SGMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Chi-Hang Lee, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRC CSA 2015
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnea; Acute Coronary Syndrome
Keywords: sleep; treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SGMT arm (Active Comparator): Treatment of OSA requires a multidisciplinary approach, involving a sleep physician and paramedical staff with expertise in the management of sleep disorders. An initial medical assessment is needed to confirm the diagnosis of OSA, determine its severity and decide whether CPAP therapy is appropriate. As part of this evaluation, an objective overnight sleep study will be performed. This will be followed by an assessment, education, and counseling at the multidisciplinary therapy clinic.
  Interventions: Device: Continuous Positive Airway Therapy; Behavioral: Sleep-Study Guided Multidisciplinary Therapy
- Control arm (No Intervention): The patients will be treated according to the standard treatment for acute coronary syndrome in Singapore, which is largely in accordance with the recommendations of the American College of Cardiology and the American Heart Association. Management includes, but is not limited to, antiplatelet and lipid-lowering therapy, early coronary revascularization, and cardiac rehabilitation, with the recommendation to follow the current practice and the most recent international guidelines.

INTERVENTIONS:
Device: Continuous Positive Airway Therapy
  Other Names: CPAP
  Arms: SGMT arm
Behavioral: Sleep-Study Guided Multidisciplinary Therapy
  Arms: SGMT arm

SUMMARY:
The aim of this randomized, open-label clinical trial is to determine the impact of Sleep Study-Guided Multidisciplinary Therapy (SGMT, i.e. continuous positive airway pressure and behavioral therapy) for obstructive sleep apnea (OSA) in the sub-acute phase of acute coronary syndrome on cardiovascular outcomes. We hypothesize that SGMT will result in a lower (1) plasma NT-pro BNP, ST2 levels and hs-CRP, (2) 10-year risk of cardiovascular mortality based on the European SCORE algorithm, and (3) cardiovascular event rate, when compared with Standard Therapy.

OSA is an emerging cardiac risk factor and prognostic marker. We have reported that OSA is a prevalent and independent predictor of adverse outcomes in patients with acute coronary syndrome. In this clinical trial, a continuation of my research and publication trajectory, 180 patients presenting with acute coronary syndrome will be randomly assigned to SGMT (n=90) or Standard Therapy (n=90) groups. Both groups will receive guideline-mandated treatment for acute coronary syndrome. Those assigned to SGMT will undergo a sleep study. Those found to have OSA will attend the SGMT clinic run by a multidisciplinary team. Advice on continuous positive airway pressure and behavioral therapy (weight loss, exercise, positional therapy, abstinence of alcohol and sleeping pills) will be given. The primary endpoint is plasma NT-pro BNP concentration at 6-month follow-up. The secondary endpoints are ST2, hs-CRP, 10-year risk of cardiovascular mortality based on the European SCORE algorithm which includes age, sex, smoking status, systolic blood pressure, and serum total cholesterol or total/HDL-cholesterol ratio. Adverse cardiovascular events at 3-year follow-up will be determined.

In our aging population with an increasing prevalence of obesity, OSA will potentially become an increasingly important contributor to cardiovascular disease. Leveraging the collective expertise of a team of cardiologists and sleep physicians, our work will benefit society by advancing our understanding of the cardiovascular benefits of screening for and treating OSA.

DETAILED DESCRIPTION:
Acute coronary syndrome is a leading cause of mortality and morbidity globally. The Principal Investigator (PI) has been conducting research on sleep medicine and cardiovascular disease since 2007. Our early work has shown that obstructive sleep apnea (OSA) is prevalent in patients presenting with an acute coronary syndrome, and carries negative prognostic implications. This Clinician Scientist Award application is centered on the potential cardiovascular benefits of a Sleep Study-Guided Multidisciplinary Therapy (SGMT) that includes continuous positive airway pressure (CPAP) and behavioral therapy for patients presenting with an acute coronary syndrome, which could lead to a potential paradigm shift in patient management during the sub-acute phase of the syndrome. For this application, we have assembled a team of experts in cardiovascular medicine and sleep medicine. Using the leverage of the synergistic expertise of the assembled leaders and the knowledge generated in the early part of the program, we will embark on a therapeutic trial.

In this randomized trial, 180 patients presenting with an acute coronary syndrome will be recruited and randomized into SGMT versus standard therapy (without sleep study) groups. Both groups will be treated with a guideline-mandated therapy for acute coronary syndrome (including regular cardiology outpatient clinic visits after discharge). In those allocated to SGMT, an overnight sleep study using a level 3 portable diagnostic device will be carried out. Those with OSA (an estimated 75% according to the pilot data) will be treated with CPAP and behavioral therapy. Plasma N-terminal pro-brain natriuretic peptide (NT-proBNP), ST2, and hs-CRP levels will be measured before hospital discharge and at 6-month follow-up. The 10-year risk of cardiovascular mortality based on the European cardiovascular risk score (SCORE), which includes age, sex, smoking status, systolic blood pressure, and serum total cholesterol or total/high-density lipoprotein (HDL)-cholesterol ratio, will be determined at baseline and at 6-month follow-up.

Our specific aims are to compare the effects of SGMT and standard therapy on:

* Plasma levels of NT-proBNP (Primary endpoint), ST2 and hs-CRP. We hypothesize that SGMT will be associated with a lower plasma NT-proBNP, ST2 and hs-CRP levels than standard therapy at 6-month follow-up.
* Systematic COronary Risk Evaluation (SCORE). We hypothesize that SGMT will be associated with a lower SCORE than standard therapy at 6-month follow-up.
* Incidence of major adverse cardiac events (extended study). We hypothesize that SGMT will be associated with a lower incidence of major adverse cardiac events at 3-year follow-up (an application for additional funding will be made to accomplish this aim).

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years, admission with an acute coronary syndrome, competent informed consent, and the ability to follow all protocol procedures.

Exclusion Criteria:

* Known OSA being treated by CPAP, recommended coronary artery bypass surgery, concomitant moderate to severe structural valve disease, clinical instability (decompensated hypotension, heart failure, shock, refractory ventricular arrhythmias, acute conduction system disease, implanted defibrillator, or left ventricular ejection fraction ≤ 30%), limited life expectancy (< 1 year) due to a concomitant illness, prior or planned heart transplant or any other organ transplant, pregnancy or current nursing activity, or inability to give informed consent.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of NT-proBNP | 6-month

SECONDARY OUTCOMES:
European cardiovascular risk SCORE | 6-month
Composite clinical endpoint of cardiovascular death, myocardial infarction (Q-wave and non-Q wave), stroke, unplanned revascularization, and hospitalization for heart failure | 12-month
Plasma concentration of ST2 | 6-month
Plasma concentration of hs-CRP | 6-month

OTHER OUTCOMES:
Compliance to CPAP | 6-month

CONTACTS AND LOCATIONS:
Locations (1):
- Chi-Hang Lee, Singapore, Singapore

REFERENCES:
- [Derived] Koo CY, Chua AP, Kristanto W, Koh EH, Tan ES, Abd Rahman S, Abd Gani MB, Chong JP, Aung AT, Han TO, Chan SP, Low AF, Yeo TC, Chan MY, Kojodjojo P, Richards AM, Lee CH. Screening and treatment of obstructive sleep apnea in acute coronary syndrome. A randomized clinical trial. Int J Cardiol. 2020 Jan 15;299:20-25. doi: 10.1016/j.ijcard.2019.07.003. Epub 2019 Jul 3. PMID 31307844